CLINICAL TRIAL: NCT01801020
Title: Different Modes of Temperature Measurement in the Emergency Department
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The investigator left the organization
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Snait Ayalon, Dr., HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMC-107-12CTIL
Record Dates: First submitted 2013-01-14; First posted 2013-02-28 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Sepsis
Keywords: temperature
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temperature measuremts (Experimental): A temporal artery measurement will be taken from two points a strait line across the forehead and an additional measurement behind the earlobe. In addition tympanic temperature will be measured.
  Interventions: Other: temperature measuremts

INTERVENTIONS:
Other: temperature measuremts — temporal artery temperature measurements will be taken from the forehead
  Other Names: LNE 0459 UTT 0537 TUV 0197 Exergen
Other: temperature measuremts — different modes of temperature measuremts will be compared to one another in the same patient. if temporal measurement is higher than oral a rectal temperature will be taken

SUMMARY:
Introduction: Temperature measurement is a crucial and integral element in the assessment of the emergency department patients. The basis of triage and treatment is often directly influenced by temperature measurement. The finding of hyper/hypothermia may differentiate between a simple urinary tract infection and pyelonephritis, or in more extreme cases may discern "weakness" in the elderly from sepsis. This brief encounter of temperature measurement may be paramount to the medical treatment of the emergency department patient. The investigators will explore the different modes of temperature measurements in emergency department patients.

DETAILED DESCRIPTION:
Temperature measurement is a crucial and integral element in the assessment of the emergency department patients. The basis of triage and treatment is often directly influenced by temperature measurement. The finding of hyper/hypothermia may differentiate between a simple urinary tract infection and pyelonephritis, or in more extreme cases may discern "weakness" in the elderly from sepsis. This brief encounter of temperature measurement may be paramount to the medical treatment of the emergency department patient.We will explore the different modes of temperature measurements in emergency department patients. We will check which temperature measurement is beneficial.

ELIGIBILITY:
Inclusion Criteria:

* patients who arrive to the emergency department

Exclusion Criteria:

* patients who refuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Different modes of temperature measurement in the emergency department | Three years
  To examine different modes of temperature measurements in emergency department patients.

SECONDARY OUTCOMES:
Different modes of temperature measurement in the emergency department | three years
  We wish to find more accurate and time efficient measurement of temperature in emergency department patients

CONTACTS AND LOCATIONS:
Overall Officials: Batshev Tzadok, MD, Principal Investigator — HaEmek Medical Center - Afula, Israel 18101
Locations (1):
- Emek Medical Center Emergency Department, Afula, Israel, Israel